CLINICAL TRIAL: NCT01964898
Title: Integrated Smoking Cessation and Mood Management for Cardiac Patients
Brief Title: Post Acute Coronary Event Smoking Study
Acronym: PACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Andrew Busch, Research Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23HL107391 (NIH)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Smoking Cessation; Acute Coronary Syndrome
Keywords: Smoking; Mood Management; Depression; Behavioral Activation; Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Smoking Cessation; Acute Coronary Syndrome; Smoking; Depression; Myocardial Infarction | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BA for cardiac patients who smoke (Experimental): Behavioral Activation Treatment for cardiac patients who smoke (BAT-CS). Participant will receive (a) 1 hour of standard smoking cessation counseling in the hospital and (b) 5 to 9 Behavioral Activation (BA) counseling sessions focused on cessation and mood management after they leave the hospital. BA sessions will occur over the 12 weeks after hospital discharge. An 8 week supply of the nicotine patch will be provided if the patient is cleared by their MD.
  Interventions: Behavioral: Behavioral Activation (BA); Behavioral: Standard Smoking Cessation Counseling; Drug: Nicotine patch
- Standard Care (Active Comparator): Participant will receive (a) 1 hour of standard smoking cessation counseling in the hospital and (b) 5 packets of printed self-help materials for smoking cessation mailed 1, 3, 6, 9, and 12 weeks after hospital discharge. An 8 week supply of the nicotine patch will be provided if the patient is cleared by their MD.
  Interventions: Behavioral: Standard Smoking Cessation Counseling; Drug: Nicotine patch; Other: Printed Self-help materials for Smoking Cessation

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) — 5 to 9 Behavioral Activation (BA) counseling sessions focused on cessation and mood management. BA sessions will occur over the 12 weeks after hospital discharge.
  Arms: BA for cardiac patients who smoke
Behavioral: Standard Smoking Cessation Counseling — 1 hour of in hospital counseling based on clinical guidelines
Drug: Nicotine patch — An 8 week supply of the nicotine patch will be provided if the patient is cleared by their MD.
Other: Printed Self-help materials for Smoking Cessation
  Arms: Standard Care

SUMMARY:
Smoking and depressed mood are both predictive of mortality following Acute Coronary Syndrome. However, to date, no counseling treatment has been designed to target smoking cessation and manage mood in this population. This trial will test such a treatment based on Behavioral Activation, an approach that has shown promise as an integrated treatment for smoking and mood management in other populations.

DETAILED DESCRIPTION:
The occurrence of Acute Coronary Syndrome (ACS; unstable angina, ST and non-ST elevation myocardial infarction) can be conceptualized as a "teachable moment," whereby patients may be more receptive to smoking cessation messages. Continued smoking following ACS is an independent predictor of mortality. Depressed mood post-ACS is also predictive of mortality, and smokers with depressed mood are less likely to abstain from smoking following an ACS hospitalization. Thus, a single, integrated treatment that targets both depressed mood and smoking could be highly effective in reducing post-ACS mortality. Behavioral Activation (BA) may be an ideal treatment for this population as BA can easily integrate both mood and smoking cessation related goals and it focuses on addressing restriction of valued activities, which is common in the post-ACS population.

Thus, the overall aim of the current study is test a BA treatment manual that integrates smoking cessation and mood management for post-ACS smokers (Behavioral Activation Treatment for cardiac patients who smoke; BAT-CS). We will conduct an RCT (N=72) comparing BAT-CS (1 in-hospital session and 5-9 post-discharge sessions) to Standard Care (SC; 1 in-hospital session and 5 mailed packets of printed self-help materials). Differences in smoking cessation, depressed mood, and positive affect will be compared between conditions.

ELIGIBILITY:
Inclusion Criteria:

* ACS diagnosis documented in medical record
* smoked 3 or more cigarettes per day before being hospitalized
* between the ages of 18-75
* fluent in English
* regular access to a telephone
* lives in the Providence, RI area
* willing to "strongly consider" an attempt to quit smoking at discharge

Exclusion criteria:

* limited mental competency (i.e., Mini-Mental Status exam < 20)
* presence of current psychosis, serious mental illness, or suicidality, expectation that patient will not live through 6 month study period
* currently regularly attending counseling for depression or smoking cessation and plans to continue after discharge

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Busch, Ph.D, Principal Investigator — The Miriam Hospital Centers for Behavioral and Preventive Medicine
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Busch AM, Tooley EM, Dunsiger S, Chattillion EA, Srour JF, Pagoto SL, Kahler CW, Borrelli B. Behavioral activation for smoking cessation and mood management following a cardiac event: results of a pilot randomized controlled trial. BMC Public Health. 2017 Apr 17;17(1):323. doi: 10.1186/s12889-017-4250-7. PMID 28415979

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 65 patients were recruited. 1 was found to be ineligible pre-randomization.
Groups:
- Standard Care: Participant will receive (a) 1 hour of standard smoking cessation counseling in the hospital and (b) 5 packets of printed self-help materials for smoking cessation mailed 1, 3, 6, 9, and 12 weeks after hospital discharge. An 8 week supply of the nicotine patch will be provided if the patient is cleared by their MD.
  Standard Smoking Cessation Counseling: 1 hour of in hospital counseling based on clinical guidelines
  Nicotine patch: An 8 week supply of the nicotine patch will be provided if the patient is cleared by their MD.
  Printed Self-help materials for Smoking Cessation
Period: Overall Study
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Started | 31 | 33
12 Week Assessment | 25 | 30
Completed (Completed assessment 6 months post-discharge) | 24 | 26
Not Completed | 7 | 7
Not completed — ineligible post-randomization | 1 | 1
Not completed — did not receive the allocated interventi | 2 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (11.9) | 57.1 (8.3) | 55.6 (10.2)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 23 | 20 | 43
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 59

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation: 7 Day Point Prevalence Abstinence
Description: No smoking, not even a puff, for 7 days; verified by carbon monoxide measurement. Results are adjusted for nicotine patch use and concurrent medication treatment targeting cessation.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
proportion of participants | 0.46 [0.28 to 0.64] | 0.44 [0.26 to 0.62]

2. Primary Outcome: Continuous Abstinence From Smoking Since Discharge
Description: Results are adjusted for nicotine patch use and concurrent medication treatment targeting cessation.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
proportion of participants | 0.38 [0.20 to 0.56] | 0.34 [0.18 to 0.50]

3. Primary Outcome: Time to Smoking Relapse
Description: Time in days to first relapse (i.e., smoking on 7 consecutive days or smoking in 2 consecutive 7 day periods), which were determined through timeline follow back interviewing. Results are adjusted for nicotine patch use and concurrent medication treatment targeting cessation.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Days
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
Days | 71.2 (17.2) | 47.4 (8.7)

4. Primary Outcome: Time to Smoking Lapse
Description: Time in days to first lapse (i.e., first puff of a cigarette) after discharge, which were determined through timeline follow back interviewing. Results are adjusted for nicotine patch use and concurrent medication treatment targeting cessation.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Days
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
Days | 62.4 (13.8) | 31.8 (6.5)

5. Secondary Outcome: Depression: 9 Item Patient Health Questionnaire (PHQ-9)
Description: The 9 item Patient Health Questionnaire (PHQ-9) ranges from 0-27 with higher scores indicating higher depression symptoms. Adjusted for anti-depressant medication use and for cardiac rehabilitation attendance.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
units on a scale
  Adjusted PHQ-9 Baseline | 6.33 (2.10) | 6.98 (1.77)
  Adjusted PHQ-9 6 months | 3.34 (2.62) | 6.08 (2.35)

6. Secondary Outcome: Depression: 10 Item Center for Epidemiologic Studies Depression Scale (CESD)
Description: The 10 item Center for Epidemiologic Studies Depression Scale ranges from 0-30 with higher scores indicating higher depression symptoms. Adjusted for anti-depressant medication use and for cardiac rehabilitation attendance.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
units on a scale
  Adjusted CESD Baseline | 10.36 (1.31) | 11.72 (1.23)
  Adjusted CESD 6 months | 5.57 (1.06) | 6.93 (1.03)

7. Secondary Outcome: Positive Affect
Description: As measured by the 10 item Positive Affect Negative Affect Scales (PANAS). The positive affect scale on the PANAS ranges from 5-25 with higher scores indicating greater positive affect in the past week. Adjusted for anti-depressant medication use and for cardiac rehabilitation attendance
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
units on a scale
  Adjusted PANAS-Positive Baseline | 13.47 (0.68) | 14.56 (0.47)
  Adjusted PANAS-Positive 6 months | 16.85 (1.66) | 15.79 (1.52)

8. Secondary Outcome: Negative Affect
Description: As measured by the 10 item Positive Affect Negative Affect Scales (PANAS). The negative affect scale on the PANAS ranges from 5-25 with higher scores indicating greater negative affect in the past week. Adjusted for anti-depressant medication use and for cardiac rehabilitation attendance.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Number analyzed (Participants) | 28 | 31
units on a scale
  Adjusted PANAS-Negative Baseline | 9.63 (0.91) | 7.62 (0.75)
  Adjusted PANAS-Negative 6 months | 7.41 (1.41) | 8.14 (0.87)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BA for Cardiac Patients Who Smoke | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No